CLINICAL TRIAL: NCT02054624
Title: Rural Lifestyle Eating and Activity Program
Brief Title: Rural Lifestyle Eating and Activity Program (Rural LEAP)
Acronym: Rural LEAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 29-2013-N; R18HL112720 (NIH); IRB201600055 (Other: UF IRB)
Record Dates: First submitted 2014-02-03; First posted 2014-02-04 (Estimated); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Obesity
Keywords: Obesity; Rural Health; Exercise; Weight loss; Behavior change
MeSH Terms: conditions — Obesity; Motor Activity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Individual (Active Comparator): The weight-loss treatments will include two phases. Phase 1 will last 4 months and Phase 2 will last 12 more months.
  Phase 1 will be 4 months of weight loss treatment
  Phase 2 will be 12 months of follow-up contact by one-on-one telephone call.
  The participants will learn about nutrition, physical activity, and safe methods to lose weight during Phase 1.
  During Phase 2 participants will receive two phone calls per month from their group leader for the first 6 months, and one phone call per month for the next 6 months.
  Interventions: Behavioral: Individual; Behavioral: All Groups
- Lifestyle intervention (Active Comparator): The weight-loss treatments will include two phases. Phase 1 will last 4 months and Phase 2 will last 12 more months.
  Phase 1 will be 4 months of weight loss treatment
  Phase 2 will be 12 months of follow-up contact by conference telephone call.
  The participants will learn about nutrition, physical activity, and safe methods to lose weight during Phase 1.
  During Phase 2 participants will receive two phone calls per month from their group leader for the first 6 months, and one phone call per month for the next 6 months.
  Interventions: Behavioral: Lifestyle intervention; Behavioral: All Groups
- Health Education Control (Active Comparator): The weight-loss treatments will include two phases. Phase 1 will last 4 months and Phase 2 will last 12 more months.
  Phase 1 will be 4 months of weight loss treatment
  Phase 2 will be 12 months of follow-up contact by email.
  The participants will learn about nutrition, physical activity, and safe methods to lose weight during Phase 1.
  During Phase 2 participants will receive a specially prepared newsletter two times per month. The newsletter will contain educational information about proper eating and physical activity. The newsletters will include low-fat and low-calorie recipes, along with tip sheets that describe strategies to help them maintain lost weight.
  Interventions: Behavioral: Health education control; Behavioral: All Groups

INTERVENTIONS:
Behavioral: Lifestyle intervention — The weight-loss treatments will include two phases. Phase 1 will last 4 months and Phase 2 will last 12 more months.
  Phase 1 will be 4 months of weight loss treatment
  Phase 2 will be 12 months of follow-up contact by group telephone call.
  The participants will learn about nutrition, physical activity, and safe methods to lose weight during Phase 1.
  During Phase 2 participants will receive two phone calls per month from their group leader for the first 6 months, and one phone call per month for the next 6 months.
  Arms: Lifestyle intervention
Behavioral: Health education control — The weight-loss treatments will include two phases. Phase 1 will last 4 months and Phase 2 will last 12 more months.
  Phase 1 will be 4 months of weight loss treatment
  Phase 2 will be 12 months of follow-up contact by email.
  The participants will learn about nutrition, physical activity, and safe methods to lose weight during Phase 1.
  During Phase 2 participants will receive a specially prepared newsletter two times per month. The newsletter will contain educational information about proper eating and physical activity. The newsletters will include low-fat and low-calorie recipes, along with tip sheets that describe strategies to help them maintain lost weight.
  Arms: Health Education Control
Behavioral: Individual — The weight-loss treatments will include two phases. Phase 1 will last 4 months and Phase 2 will last 12 more months.
  Phase 1 will be 4 months of weight loss treatment
  Phase 2 will be 12 months of follow-up contact by on-on-one telephone call.
  The participants will learn about nutrition, physical activity, and safe methods to lose weight during Phase 1.
  During Phase 2 participants will receive two phone calls per month from their group leader for the first 6 months, and one phone call per month for the next 6 months.
  Arms: Individual
Behavioral: All Groups — All participants will receive the following: Questionnaires, height, weight, waist measurement, blood pressure, heart rate, electrocardiogram, blood sample, urine sample, urine pregnancy test (for females only), 400 meter walking test

SUMMARY:
The purpose of this research study is to learn about ways to help adults with obesity from rural areas manage their weight and increase their physical activity. An important goal of the study is to find out what type of follow-up program for weight management is necessary to help adults with obesity keep from regaining lost weight. The study will also look at the ways that long-term weight-loss treatments affect blood pressure, blood fats (lipids), blood sugar, and physical fitness.

The participant are being asked to be in this research study because increased weight and obesity are major health problems in the United States. The participant's weight and height fall in the obese category. Adults with obesity have an increased risk of developing health problems such as high blood pressure, diabetes, and heart disease. The rates of being overweight and obese are higher in rural areas of the United States than in urban and suburban areas of the country.

DETAILED DESCRIPTION:
If the participant agrees to participate, a number of tests will be performed to see if the participant is eligible to take part in the study. If so, these tests will be repeated after 4 months of treatment, and again after 22 months. Participants will be asked to complete a number of questionnaires. baseline, 4 months of treatment, and again after 10, 16, and 22 months. The different tests and measures are listed below.

Questionnaires, Height, Weight, Waist Measurement, Blood Pressure, Heart Rate, Electrocardiogram, Blood Sample (2 tablespoons), Urine Sample, and a Urine Pregnancy test for females, 400 Meter Walking Test

Randomization

A member of the research team will contact participants by telephone or by mail if they eligible to take part in the study. Participants are randomly assigned to one of three groups. Random assignment is like rolling dice to decide which group a person is assigned to.

The three groups are described below:

Group A: 4 months of weight loss treatment plus 12 months of follow-up contact by telephone. The follow-up telephone contacts in Group A will involve group discussion with a trained staff member and other participants.

Group B: 4 months of weight loss treatment plus 12 months of follow-up contacts by telephone. The follow-up telephone contacts in Group B will involve individual, one-on-one discussion with a trained staff member.

Group C: 4 months of weight loss treatment plus 12 months of follow-up contacts by mail and e-mail.

Weight Loss Treatments

The weight-loss treatments in this study will include two phases. Phase 1 will last 4 months. Phase 2 will last 12 more months. Everybody in Groups A, B, and C will have the same Phase 1 weight-loss treatment program for 4 months. However, the type of Phase 2 follow-up program that participants receive will depend on whether they are assigned to Group A, B, or C.

Phase 1 Treatment

During this time, participants will meet each week with a group leader and a group of about 10 other adults. The meetings will take place at the Cooperative Extension Office. The group leader will be a Family and Consumer Sciences Agent who has had special training in nutrition education or a staff member who has had special training in weight-management. The group meetings will last about 90 minutes per week. All group meeting will be audio recorded so that the researchers can determine if the treatment was delivered as planned.

There are four major goals for the group sessions.

1. Participants will learn about nutrition, physical activity, and safe methods to lose weight. To help accomplish this goal, participants will be asked to keep a daily habit log on which participants will record everything they eat and drink each day. Participants will also be given a pedometer. A pedometer is a small device about the size of a pager that keeps track of how many steps the participant takes each day. Participants will be asked to wear the pedometer each day, and write down on thier habit log each day the number of steps tracked by thier pedometer.
2. Participants will be taught how to eat a healthy diet while taking in fewer calories than they are currently eating. This will usually mean reducing calorie intake by 500 to 1000 calories per day. Participants will participate in cooking demonstrations and will have a chance to sample healthy foods prepared during group meetings.
3. Participants will be taught how to set up a regular routine of increased physical activity or exercise. This will usually involve a walking program of 30 minutes per day.
4. Participants will be taught ways to increase their motivation to start and maintain changes in their eating and exercise habits.

Phase 2 Treatments

Phase 2 of the program will begin after the completion of Phase 1 and will last for 12 months. Phase 2 will involve follow-up programs to help group members continue their weight management efforts. During Phase 2 participants will be encouraged to maintain improved, healthy patterns of exercise and dietary intake, and to continue to monitor and record their dietary intake and pedometer steps on a regular basis.

The follow-up programs for all Groups will involve two contacts per month for the first 6 months and one contact per month for the next 6 months. However, the type of contact will be different for each Treatment Group.

Group A: This group will have follow-up contact by phone. If participants are assigned by the computer to Group A, they will receive two phone calls per month from their group leader for the first 6 months, and one phone call per month for the next 6 months. These calls will be group phone calls; other participants will be on the call. These group phone calls will be led by a trained group leader and will include discussions of progress and will focus on strategies to help participants maintain lost weight.

Group B: This group will have follow-up contact by phone. If participants are assigned by the computer to Group B, they will receive two phone calls per month from their group leader for the first 6 months, and one phone call per month for the next 6 months. These calls will be individual phone calls with the participant and a trained staff member that will include discussions of progress and will focus on strategies to help them maintain lost weight.

Group C: This group will have follow-up contact by mail. If participants are assigned by the computer to Group C, they will receive a specially prepared newsletter two times per month. The newsletter will contain educational information about proper eating and physical activity. The newsletters will include low-fat and low-calorie recipes, along with tip sheets that describe strategies to help them maintain lost weight.

If participants are in Group A or B four of their phone call treatment sessions will be audio recorded so that the researchers can determine if the treatment was delivered as planned.

ELIGIBILITY:
Inclusion Criteria:

* Age: 21 to 75 years
* Body Mass Index: 30 to 45 kg/m**2

Exclusion Criteria:

* Underlying disease likely to limit lifespan and/or increase risk of interventions:cancer requiring treatment in past five years (exception: non-melanoma skin cancer); serious infectious diseases (e.g., self-reported HIV, self-reported tuberculosis or treatment); myocardial infarction or cerebrovascular accident within the last six months; unstable angina within the past six months; congestive heart failure; chronic hepatitis; cirrhosis; chronic malabsorption syndrome; chronic pancreatitis; irritable bowel syndrome; previous bariatric surgery; history of organ transplantation; history of musculoskeletal conditions that limit walking; chronic lung diseases that limit physical activity; and any other condition likely to limit five-year life expectancy.
* Metabolic exclusions: fasting blood glucose > 125 mg/dl at screening if not known to be diabetic (patients with diabetes under active treatment will be enrolled if approved by primary provider); fasting serum triglycerides > 400 mg/dl at screening; resting blood pressure > 150/100 mm Hg.
* Medication exclusions: antipsychotic agents; monoamine oxidase inhibitors; systemic corticosteroids; antibiotics for HIV or Tuberculosis; chemotherapeutic drugs; or use of prescription weight-loss drugs within six months.
* Conditions or behaviors likely to affect the conduct of the trial: unwilling or unable to give informed consent; unable to read English at the 5th grade level; unwilling to accept random assignment; unwilling to travel to Extension office for intervention sessions; participation in another randomized research project; weight loss > 10 pounds in past six months; likely to move out of the county in next two years; major psychiatric disorder; excessive alcohol intake; BMI > 45; prior participation in the TOURS trial; and other conditions which in the opinion of staff would adversely affect participation in the trial

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 631 (Actual)
Dates: Start 2013-08; Primary Completion 2018-12 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Change in body weight (kg) from month 4 to month 22 | Change from month 4 to month 22
  Weight is measured on a Tanita digital scale.

SECONDARY OUTCOMES:
Percent of participants achieving 5% or greater weight losses at month 22 | Baseline to month 22
  Weight is measured on a Tanita digital scale.
Percent of participants achieving 10% or greater weight losses at month 22 | Baseline to month 22
  Weight is measured on a Tanita digital scale.

OTHER OUTCOMES:
Blood pressure (mmHg) from baseline to month 4 | Change from baseline to month 4
  A clinical staff member will take the blood pressure from the right arm and also count the heart rate for 30 seconds. Blood pressure and heart rate will be measured 1 or 2 more times. The change in systolic and diastolic blood pressure from baseline to four months will be reported.
LDL-Cholesterol (mg/dL) change in baseline to month 4 | Change from baseline to month 4
  A staff member will take about 2 tablespoons of blood from the arm. The blood will be studied to find out the levels of LDL-Cholesterol concentration in blood.
HDL-Cholesterol (mg/dL) change in baseline to month 4 | Change from baseline to month 4
  A staff member will take about 2 tablespoons of blood from the arm. The blood will be studied to find out the levels of HDL-Cholesterol concentration in blood.
Triglycerides (mg/dL) change from baseline to month 4 | Change from baseline to month 4
  A staff member will take about 2 tablespoons of blood from the arm. The blood will be studied to find out the levels of triglyceride concentration in blood.
Fasting blood glucose (mmol/L) change in baseline to month 4 | Change from baseline to month 4
  A staff member will take about 2 tablespoons of blood from the arm. The blood will be studied to find out the levels of fasting blood glucose in blood.
Glycated hemoglobin (hemoglobin A1c, HbA1c, A1c) | Change in glycated hemoglobin from baseline to month 4
  A staff member will take about 2 tablespoons of blood from the arm. The blood will be studied to find out the levels of sugar the blood.
400 meter walk test (m/s) | Change in pace from baseline to four months
  A trained staff member will supervise participants in the completion of a 400 Meter walking test. They will be instructed to walk 400 meters at a standard pace on a clearly marked indoor course. Time it takes to complete the walk will be recorded. Participants will be allowed to stop and rest or stop and not complete the test at anytime.
Physical activity - steps | Change in average daily step count from baseline to four months
  A pedometer will be worn on the waist to record the number of steps taken each day.
Dietary intake (kcals) | Change in caloric intake from baseline to four months
  Daily habit logs will be kept including details on all foods and beverage eaten each day. Specifically, name of food/beverage, amount and calorie content will be recorded.
Dietary intake | Change in caloric intake from baseline to four months
  This questionnaire asks questions about participants overall dietary intake over the last year.
Waist circumference (cm) | Change in waist circumference from baseline to four months
  A staff member will use a tape measure to measure participants waist.
Health Related Quality of Life | Change in Health Related Quality of Life measured by Likert scale from baseline to month four
  These questionnaires ask about health, eating and exercise habits, and thoughts and feelings. This information will be used to help determine how personal factors (e.g., age, gender, race, education, income, marital status) are associated with change in weight.
Cost Analysis | Cost effectiveness of the intervention from baseline to month four
  Questionnaires asking about background information will be completed to assess the economic impact of this program.
Blood pressure (mmHg) | Change in systolic and diastolic blood pressure from baseline to 22 months
  Participants will sit quietly for 5 minutes without talking or distractions. The clinical staff member will then take their blood pressure from the right arm. The staff member will also count the heart rate for 30 seconds. Participants blood pressure and heart rate will be measured 1 or 2 more times.
LDL-Cholesterol (mg/dL) | Change in blood LDL-Cholesterol concentration from baseline to 22 months
  The staff member will take about 2 tablespoons of blood from participants arm. The blood will be studied to find out the levels of fats (lipids) in the blood.
HDL-Cholesterol (mg/dL) | Change in blood HDL-Cholesterol concentration from baseline to 22 months
  The staff member will take about 2 tablespoons of blood to find out the levels of fats (lipids) in participants blood.
Triglycerides (mg/dL) | Change in blood triglyceride concentration from baseling to 22 months
  The blood will be studied to find out the levels of fats (lipids) in the participants blood.
Fasting blood glucose (mmol/L) | Change in fasting blood glucose concentration from baseline to 22 months
  The blood will be studied to find out the levels of sugar in the participants blood.
Glycated hemoglobin (hemoglobin A1c, HbA1c, A1c) | Change in glycated hemoglobin from baseline to month 22
  The blood will be studied to find out the levels of sugar in the participants blood.
400 meter walk test (m/s) | Change in pace from baseline to 22 months
  A trained staff member will supervise participants in the completion of a 400 Meter walking test. Participants will be instructed to walk 400 meters at their own pace, and the time it takes them to complete the walk will be recorded. Participants will walk on a clearly marked indoor course. They will be allowed to stop and rest or stop and not complete the test at anytime. If they experience any abnormal symptoms during the test, such as chest pain or severe shortness of breath, they should immediately inform the test supervisor. If they experience any symptoms during the walk, such as shortness of breath, feelings of dizziness, or excessive tiredness (fatigue), they will be asked to remain in the testing area for 15 minutes of observation following the test.
Physical activity - steps | Change in average daily step count from baseline to 22 months
  Participants will be given a pedometer (at no cost to them). A pedometer is a small device about the size of a pager that keeps track of how many steps are taken each day. Participants will be asked to wear the pedometer each day, and write down on their habit log each day the number of steps tracked by their pedometer.
Dietary intake (kcals) | Change in caloric intake from baseline to 22 months
  Participants will be asked to keep a daily habit log on which they will record everything they eat and drink each day. Specifically, name of food/beverage, amount and calorie content will be recorded.
Dietary intake | Change in caloric intake from baseline to 22 months
  This questionnaire asks questions about their overall dietary intake over the last year.
Waist circumference (cm) | Change in waist circumference from baseline to 22 months
  A staff member will use a tape measure to measure their waist.
Health Related Quality of Life | Change in Health Related Quality of Life measured by Likert scale from baseline to month 22
  Participants will be asked to fill out some questionnaires that ask about health, eating and exercise habits, and their thoughts and feelings. This information will be used to help us understand how personal factors (e.g., age, gender, race, education, income, marital status) are associated with change in weight.
Cost Analysis | Cost effectiveness of the intervention from baseline to month 22
  Participants will be asked to complete a background information questionnaire; this information will be used to assess the economic impact of this program.

CONTACTS AND LOCATIONS:
Overall Officials: Michael G Perri, Ph.D., ABPP, Principal Investigator — University of Florida
Locations (14):
- United States (14):
  - Levy County, Bronson, Florida
  - Flagler County, Bunnell, Florida
  - Dixie County, Cross City, Florida
  - Hamilton County, Jasper, Florida
  - Union County, Lake Butler, Florida
  - Columbia County, Lake City, Florida
  - Suwannee County, Live Oak, Florida
  - Baker County, Macclenny, Florida
  - Madison County, Madison, Florida
  - Lafayette County, Mayo, Florida
  - Putnam County, Palatka, Florida
  - Taylor County, Perry, Florida
  - Bradford County, Starke, Florida
  - Gilchrist County, Trenton, Florida

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Perri MG, Shankar MN, Daniels MJ, Durning PE, Ross KM, Limacher MC, Janicke DM, Martin AD, Dhara K, Bobroff LB, Radcliff TA, Befort CA. Effect of Telehealth Extended Care for Maintenance of Weight Loss in Rural US Communities: A Randomized Clinical Trial. JAMA Netw Open. 2020 Jun 1;3(6):e206764. doi: 10.1001/jamanetworkopen.2020.6764. PMID 32539150
- [Derived] Perri MG, Ariel-Donges AH, Shankar MN, Limacher MC, Daniels MJ, Janicke DM, Ross KM, Bobroff LB, Martin AD, Radcliff TA, Befort CA. Design of the Rural LEAP randomized trial: An evaluation of extended-care programs for weight management delivered via group or individual telephone counseling. Contemp Clin Trials. 2019 Jan;76:55-63. doi: 10.1016/j.cct.2018.11.006. Epub 2018 Nov 6. PMID 30408606
- See also: Design of the Rural LEAP randomized trial: An evaluation of extended-care programs for weight management delivered via group or individual telephone counseling — https://doi.org/10.1016/j.cct.2018.11.006